CLINICAL TRIAL: NCT00406341
Title: Phase 3 Confimatory Study of 0.05% Difluprednate Ophthalmic Emulsion in the Treament of Postoperative Inflammation
Brief Title: Study of Difluprednate Ophthalmic Emulsion in Postoperative Inflammation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sirion Therapeutics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SJE2079/3-03
Record Dates: First submitted 2006-11-29; First posted 2006-12-04 (Estimated); Last update posted 2006-12-04 (Estimated); Status verified 2006-11

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation

INTERVENTIONS:
Drug: Difluprednate Ophthalmic Emulsion

SUMMARY:
The purpose of this phase 3 study is to determine if difluprednate ophthalmic emulsion is effective in the treatment of postoperative inflammation.

DETAILED DESCRIPTION:
The objective of this phase 3 study is to assess the efficacy and safety of 0.05% difluprednate ophthalmic emulsion in patients with intraocular postoperative inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone cataract surgery, vitreous surgery or both (including patients who have undergone IOL insertion surgery at the same time)
* Patients showing an anterior chamber cell score of not less than "2" at a day after surgery
* Patients aged 20 years or over, irrespective of genders (it is eligible for enrollment when patients' age attains the criterion on the day of consent obtainment)

Exclusion Criteria:

* Patients who took systemic administration of corticosteroids or immunosuppressive agents, or used ophthalmic ointments of corticosteroids within 1 week before instillation of the investigational drugs;
* Patients who underwent local injection of corticosteroids in the eyes before instillation of the investigational drugs; (patients who used aqueous preparations within 1 week or patient who used depot preparations within 2 weeks were excluded)
* Patients who took systemic administration of non-steroidal antiinflammatory agents or antiinflammatory enzyme preparations within 3 days before instillation of the investigational drugs;
* Patients who instilled of corticosteroids, no-steroidal antiinflammatory agents or antiinflammatory enzyme preparations within 24 hours before the pre-instillation observation (a day after surgery);
* Patients who underwent perioperative and/or postoperative intravitreous injection of corticosteroids;
* Patients who underwent sub-conjunctival injection or sub-Tenon capsule injection of corticosteroids;
* Patients who have intraocular hemorrhage with a degree that may affect the postoperative evaluations;
* Patients who underwent gas tamponade at the surgery;
* Patients with endogenous uveitis;
* Patients having corneal epithelial detachment or corneal ulcer in the target eye;
* Patients who are suspected of having viral, bacterial or mycotic keratoconjunctival disorders in the target or opposite eye;
* Patients with glaucoma or ocular hypertension, or those with past history of IOP increased due to instillation of corticosteroids, or those whose IOP has been controlled by use of ophthalmic antihypertensive agents;
* Patients showing IOP not less than 25 mmHg a day after surgery;
* Patients who have allergy to corticosteroid drugs;
* Patients who are required to wear contact lens during the study period;
* Patients who are scheduled to undergo surgery of the opposite eye during the study period;
* Patients who are pregnant or may be pregnant or lactating;
* Patients who have participated in other clinical studies within 3 months.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2004-04; Study Completion 2005-03

PRIMARY OUTCOMES:
The changes in anterior chamber cell score at day 14 after start of instillation from the baseline level (differences from the baseline score) were compared between the 2 treatment groups.

SECONDARY OUTCOMES:
The changes in anterior chamber cell score at days 3 and 7 after start of instillation were compared between the 2 treatment groups.
The numbers of patients showing an anterior chamber cell score of "0" at days 3, 7 and 14 after start of instillation were compared between the 2 treatment groups.
The changes in anterior chamber flare score at days 3, 7 and 14 after start of instillation (difference from the baseline score) were compared between the 2 treatment groups.
The changes in the total scores of subjective symptoms and objective signs at days 3, 7 and 14 after start of instillation (difference from the baseline score) were compared between the 2 treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Shigeaki Ohno, Study Chair — Department of Ophthalmology and Visual Sciences, Graduate School of Medicine, Hokkaido University